CLINICAL TRIAL: NCT02552212
Title: Phase 3, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate Efficacy and Safety of Certolizumab Pegol in Subjects With Active Axial Spondyloarthritis (axSpA) Without X-Ray Evidence of Ankylosing Spondylitis (AS) and Objective Signs of Inflammation
Brief Title: Multicenter Study Evaluating Certolizumab Pegol Compared to Placebo in Subjects With axSpA Without X-ray Evidence of AS
Acronym: C-AXSPAND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS0006; 2015-001894-41 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Axial Spondyloarthritis; Nonradiographic Axial Spondyloarthritis; Nr-axSpA
Keywords: Axial Spondyloarthritis; axSpA; Ankylosing Spondylitis; Anti TNF-alpha; Certolizumab Pegol; Nr-axSpA; Non-radiographic; Spondylarthropathies; Arthritis; Spinal Diseases; Immunosuppressive Agents
MeSH Terms: conditions — Axial Spondyloarthritis; Non-Radiographic Axial Spondyloarthritis; Spondylitis, Ankylosing; Spondylarthropathies; Arthritis; Spinal Diseases | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Certolizumab Pegol 200 mg Q2W (Experimental): Certolizumab Pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 6 onwards.
  Interventions: Biological: Certolizumab Pegol
- Placebo (Placebo Comparator): Matching placebo to Certolizumab Pegol (CZP) injections are administered every 2 weeks from Week 0 onwards.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Certolizumab Pegol — * Active Substance: Certolizumab Pegol
  * Pharmaceutical Form: Prefilled syringe
  * Concentration: 200 mg / ml
  * Route of Administration: Subcutaneous injection
  Other Names: Cimzia; CDP870
  Arms: Certolizumab Pegol 200 mg Q2W
Other: Placebo — * Active Substance: Placebo
  * Pharmaceutical Form: Prefilled syringe
  * Concentration: 0.9 % saline
  * Route of Administration: Subcutaneous injection
  Arms: Placebo

SUMMARY:
Patients with active Axial Spondyloarthritis without x-ray evidence of Ankylosing Spondylitis and with signs of inflammation will be randomly assigned to receive certolizumab pegol (CZP) 200 mg every two weeks or placebo. The primary objective is to demonstrate the efficacy of CZP in these patients.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old at the start of Screening Visit
* A documented diagnosis of adult-onset axial SpondyloArthritis (axSpA) and meet the Assessment of SpondyloArthritis International Society (ASAS) criteria for axSpA
* Subjects must have had back pain for at least 12 months before Screening
* No sacroiliitis defined by Modified New York (mNY) criteria on sacroiliac (SI) x-rays
* Active disease at Screening as defined by

  * Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score >= 4
  * Spinal pain >= 4 on a 0 to 10 Numerical Rating Scale (NRS)
* Inadequate response to, have a contraindication to, or have been intolerant to at least 2 Nonsteroidal Anti-Inflammatory Drugs (NSAIDs)

Exclusion Criteria:

* Diagnosis of AS or any other Inflammatory Arthritis
* Prior treatment with any experimental biological agents for treatment of Axial SpondyloArthritis (SpA)
* Exposure to more than 1 tumor necrosis factor (TNF)-antagonist or primary failure to TNF antagonist therapy
* History of or current chronic or recurrent infections
* Subjects with known Tuberculosis (TB) infection, at high risk of acquiring TB infection, or latent Tuberculosis (LTB)
* Recent live vaccination
* Concurrent malignancy or a history of malignancy
* Class III or IV congestive heart failure - New York Heart Association (NYHA)
* Demyelinating disease of the central nervous system
* Female subjects who are breastfeeding, pregnant or plan to become pregnant during the study or within 3 months following the last dose of the investigational product
* Subjects with any other condition which, in the investigator's judgment, would make the subject unsuitable for inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 1-844-599-2273 (UCB)
Locations (105):
- United States (36):
  - As0006 125, Birmingham, Alabama
  - As0006 120, Scottsdale, Arizona
  - As0006 115, Tucson, Arizona
  - As0006 155, Beverly Hills, California
  - As0006 101, Palm Desert, California
  - As0006 143, San Francisco, California
  - As0006 160, New Haven, Connecticut
  - As0006 117, Daytona Beach, Florida
  - As0006 116, DeBary, Florida
  - As0006 124, Fort Lauderdale, Florida
  - As0006 133, New Port Richey, Florida
  - As0006 138, Plantation, Florida
  - As0006 134, Tampa, Florida
  - As0006 106, Vero Beach, Florida
  - As0006 148, Atlanta, Georgia
  - As0006 137, Idaho Falls, Idaho
  - As0006 102, Cumberland, Maryland
  - As0006 141, Cumberland, Maryland
  - As0006 111, Wheaton, Maryland
  - As0006 127, Boston, Massachusetts
  - As0006 147, Worcester, Massachusetts
  - As0006 110, Eagan, Minnesota
  - As0006 123, Rochester, Minnesota
  - As0006 103, St Louis, Missouri
  - As0006 114, Brooklyn, New York
  - As0006 118, Charlotte, North Carolina
  - As0006 149, Oklahoma City, Oklahoma
  - As0006 105, Portland, Oregon
  - As0006 108, Duncansville, Pennsylvania
  - As0006 144, Philadelphia, Pennsylvania
  - As0006 129, Wyomissing, Pennsylvania
  - As0006 156, Orangeburg, South Carolina
  - As0006 107, Salt Lake City, Utah
  - As0006 104, Seattle, Washington
  - As0006 158, Manitowoc, Wisconsin
  - As0006 113, Onalaska, Wisconsin
- Australia (7):
  - As0006 208, Camperdown
  - As0006 210, Coffs Harbour
  - As0006 204, Footscray
  - As0006 201, Malvern East
  - As0006 209, Maroochydore
  - As0006 205, South Hobart
  - As0006 202, Victoria Park
- Bulgaria (8):
  - As0006 302, Plovdiv
  - As0006 305, Plovdiv
  - As0006 304, Rousse
  - As0006 306, Sevlievo
  - As0006 300, Sofia
  - As0006 307, Sofia
  - As0006 309, Sofia
  - As0006 308, Varna
- Canada (2):
  - As0006 152, Edmonton
  - As0006 150, Victoria
- Czechia (12):
  - As0006 326, Hlučín
  - As0006 324, Hustopeče
  - As0006 327, Olomouc
  - As0006 320, Ostrava
  - As0006 322, Pardubice
  - As0006 323, Prague
  - As0006 328, Prague
  - As0006 329, Prague
  - As0006 330, Prague
  - As0006 333, Příbor
  - As0006 332, Rychnov nad Kněžnou
  - As0006 331, Zlín
- Hungary (4):
  - As0006 365, Balatonfüred
  - As0006 362, Budapest
  - As0006 363, Budapest
  - As0006 361, Székesfehérvár
- Poland (14):
  - As0006 406, Bydgoszcz
  - As0006 400, Elblag
  - As0006 401, Krakow
  - As0006 402, Krakow
  - As0006 411, Lublin
  - As0006 403, Poznan
  - As0006 404, Poznan
  - As0006 405, Torun
  - As0006 407, Warsaw
  - As0006 408, Warsaw
  - As0006 409, Warsaw
  - As0006 410, Warsaw
  - As0006 413, Wroclaw
  - As0006 414, Wroclaw
- Russia (18):
  - As0006 461, Chelyabinsk
  - As0006 453, Ivanovo
  - As0006 450, Kazan'
  - As0006 451, Kazan'
  - As0006 458, Kemerovo
  - As0006 455, Moscow
  - As0006 466, Moscow
  - As0006 462, Orenburg
  - As0006 452, Ryazan
  - As0006 459, Saint Petersburg
  - As0006 463, Saint Petersburg
  - As0006 464, Saint Petersburg
  - As0006 467, Saint Petersburg
  - As0006 465, Samara
  - As0006 454, Saratov
  - As0006 460, Smolensk
  - As0006 456, Tolyatti
  - As0006 457, Yaroslavl
- Taiwan (4):
  - As0006 232, Hualien City
  - As0006 230, Taichung
  - As0006 233, Taichung
  - As0006 231, Taipei

REFERENCES:
- [Result] van der Heijde D, Gensler LS, Maksymowych WP, Landewe R, Rudwaleit M, Bauer L, Kumke T, Kim M, Auteri SE, Hoepken B, Deodhar A. Long-term safety and clinical outcomes of certolizumab pegol treatment in patients with active non-radiographic axial spondyloarthritis: 3-year results from the phase 3 C-axSpAnd study. RMD Open. 2022 Mar;8(1):e002138. doi: 10.1136/rmdopen-2021-002138. PMID 35296532
- [Result] Robinson PC, Maksymowych WP, Gensler LS, Hall S, Rudwaleit M, Hoepken B, Bauer L, Kumke T, Kim M, de Peyrecave N, Deodhar A. Certolizumab Pegol Efficacy in Patients With Non-Radiographic Axial Spondyloarthritis Stratified by Baseline MRI and C-Reactive Protein Status: An Analysis From the C-axSpAnd Study. ACR Open Rheumatol. 2022 Sep;4(9):794-801. doi: 10.1002/acr2.11469. Epub 2022 Jun 22. PMID 35733363
- [Derived] Maksymowych WP, Kumke T, Auteri SE, Hoepken B, Bauer L, Rudwaleit M. Predictors of long-term clinical response in patients with non-radiographic axial spondyloarthritis receiving certolizumab pegol. Arthritis Res Ther. 2021 Oct 29;23(1):274. doi: 10.1186/s13075-021-02650-4. PMID 34715908
- [Derived] Deodhar A, Gensler LS, Kay J, Maksymowych WP, Haroon N, Landewe R, Rudwaleit M, Hall S, Bauer L, Hoepken B, de Peyrecave N, Kilgallen B, van der Heijde D. A Fifty-Two-Week, Randomized, Placebo-Controlled Trial of Certolizumab Pegol in Nonradiographic Axial Spondyloarthritis. Arthritis Rheumatol. 2019 Jul;71(7):1101-1111. doi: 10.1002/art.40866. Epub 2019 May 28. PMID 30848558
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll participants in September 2015. The study included a Screening Period, up to 6 weeks before Baseline, a Double-Blind (DB) Period from Baseline (Week 0) to Week 52, that included the open label CZP (OL-CZP) treatment and other treatment (OT) and an Open Label Safety Follow-up Extension (SFE) Period, up to Week 156.
Pre-assignment Details: The Participant Flow refers to the Randomized Set (RS).
Groups:
- Placebo: Matching placebo to certolizumab pegol (CZP) injections were administered every 2 weeks from Week 0 onwards.
- CZP 200 mg Q2W: Certolizumab pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 6 onwards.
- SFE OL CZP 200 mg Q2W: Subjects who completed Double-Blind Period received CZP 200 mg at Week 52, 54 and 56 to maintain the blinding and who completed the Week 52 Visit on placebo treatment received loading doses of CZP 400 mg at these visits. Subjects who completed the Week 52 Visit on CZP treatment received 1 injection of CZP 200 mg and 1 injection of placebo at these visits to continue their previous CZP treatment regimen and subjects who discontinued from Double-Blind Period and entered OL CZP treatment continued their OL CZP treatment regimen during Safety Follow-Up Extension (SFE) Period. Subjects received CZP 200 mg Q2W for up to 2 years during the SFE Period. An additional signed informed consent for the SFE was a pre-requisite For the additional milestone one (Received OL CZP; Completed Week 52 without starting SFE) reported in Double-Blind Period (Week 0 -52).
Period: Double-Blind Period (Week 0 - 52)
Arm/Group | Placebo | CZP 200 mg Q2W | SFE OL CZP 200 mg Q2W
Started | 158 | 159 | 0
Received OL CZP | 96 | 20 | 0
Completed Week 52 Without Starting SFE | 20 | 22 | 0
Completed | 143 | 142 | 0
Not Completed | 15 | 17 | 0
Not completed — Adverse Event | 6 | 3 | 0
Not completed — Lack of Efficacy | 2 | 2 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 7 | 0
Not completed — Study non-compliance | 1 | 1 | 0
Not completed — Patient's decision | 0 | 1 | 0
Not completed — As per suggestion | 0 | 1 | 0
Not completed — Not eligible | 0 | 1 | 0
Not completed — Missing/Unspecified | 1 | 0 | 0
Period: SFE Period (Week 52 - 156)
Arm/Group | Placebo | CZP 200 mg Q2W | SFE OL CZP 200 mg Q2W
Started | 0 | 0 | 243 (123 subjects from Placebo arm and 120 subjects from CZP 200 mg Q2W arm)
Completed | 0 | 0 | 206
Not Completed | 0 | 0 | 37
Not completed — Adverse Event | 0 | 0 | 5
Not completed — Lack of Efficacy | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 18
Not completed — Return to standard-of-care /OL CZP | 0 | 0 | 1
Not completed — Patient's personal reason | 0 | 0 | 1
Not completed — Investigator decision | 0 | 0 | 1
Not completed — Subject withdrew consent due to traveling to site | 0 | 0 | 1
Not completed — Compassionate access | 0 | 0 | 2
Not completed — Patient travelling for study unable to continue | 0 | 0 | 1
Not completed — Decision of Patient | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set witch consisted of all subjects randomized into the study.
Arm/Group | Placebo | CZP 200 mg Q2W | Total Title
Number analyzed (Participants) | 158 | 159 | 317
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 4
  Between 18 and 65 years | 154 | 156 | 310
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (10.8) | 37.3 (10.5) | 37.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 81 | 163
  Male | 76 | 78 | 154
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8 | 5 | 13
  Black | 1 | 0 | 1
  White | 148 | 152 | 300
  Other/mixed | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Ankylosing Spondylitis Disease Activity Score Major Improvement (ASDAS-MI) Response Criteria Response at Week 52
Description: This variable was considered as primary in all countries except for Canada (and any other country where applicable or where requested by Regulatory Authorities) where it was considered as secondary variable.
  ASDAS-MI was achieved when there was a reduction (improvement) >= 2.0 in the ASDAS relative to Baseline, or when the lowest possible ASDAS score (0.6) was reached.
  The ASDAS was calculated as the sum of the following components:
  0.121 × Back pain (BASDAI Q2 result) 0.058 × Duration of morning stiffness (BASDAI Q6 result) 0.110 × Patient's Global Assessment of Disease Activity (PGADA) 0.073 × Peripheral pain/swelling (BASDAI Q3 result) 0.579 × (natural logarithm [ln] of the (CRP [mg/L] + 1)) Back pain, PGADA, duration of morning stiffness, peripheral pain/swelling and fatigue were all assessed on a numerical scale (0 to 10 units, where 0 is "not active" and 10 is "very active").
Time Frame: Week 52
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Number; unit: percentage of subjects
Groups:
- Placebo (FAS): Matching placebo to certolizumab pegol (CZP) injections were administered every 2 weeks from Week 0 onwards. Subjects formed the Full Analysis Set (FAS).
- CZP 200 mg Q2W (FAS): Certolizumab pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 6 onwards. Subjects formed the FAS.
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 159
percentage of subjects | 7.0 | 47.2
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); Odds ratio: CZP/Placebo and p-value were calculated using logistic regression with factors for treatment, region and Magnetic Resonance Imaging/C- Reactive Protein (MRI/CRP) classification; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 15.231, 95% CI 2-sided [7.336 to 31.623]

2. Primary Outcome: Percentage of Subjects With Axial SpondyloArthritis International Society 40% Response Criteria (ASAS40) Response at Week 12
Description: This variable was considered as primary for Canada (and any other country where applicable or where requested by Regulatory Authorities) and as secondary variable in all other countries.
  The ASAS40 response was defined as relative improvements of at least 40 % and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS), where 0 is "not active" and 10 is "very active" in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)) questions 5 and 6 concerning morning stiffness intensity and duration) and no worsening at all in the remaining domain.
Time Frame: Week 12
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 159
percentage of subjects | 11.4 | 47.8
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); Odds ratio: CZP/Placebo and p-value were calculated using logistic regression with factors for treatment, region and MRI/CRP classification; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.436, 95% CI 2-sided [4.127 to 13.401]

3. Primary Outcome: Certolizumab Pegol Plasma Concentration at Baseline
Description: Certolizumab pegol plasma concentration was measured at Baseline in micrograms per millilitre (µg/mL).
Time Frame: Baseline (Week 0)
Population: The Safety Set (SS) consisted of all subjects who have received at least 1 dose of study medication. Note: None of the Safety Set subjects had Pharmacokinetic (PK) concentrations above the lower limit of quantification.
Groups:
- Placebo (SS): Matching placebo to certolizumab pegol (CZP) injections were administered every 2 weeks from Week 0 onwards. Subjects formed the Safety Set (SS).
- CZP 200 mg Q2W (SS): Certolizumab pegol (CZP) 400 mg subcutaneous (sc) on Weeks 0, 2 and 4, followed by 200 mg CZP sc every 2 weeks (Q2W) from Week 6 onwards. Subjects formed the SS.
Arm/Group | Placebo (SS) | CZP 200 mg Q2W (SS)
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Certolizumab Pegol Plasma Concentration at Week 1
Description: Certolizumab pegol plasma concentration was measured at Week 1, in µg/mL.
Time Frame: Week 1
Population: The SS consisted of all subjects who received at least 1 dose of study treatment. Note: No samples taken at Week 1 for the Placebo->OL CZP.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Groups:
- Placebo->OL CZP (SS): Subset of subjects from the Placebo group, who discontinued the CZP double-blind treatment and entered the open-label CZP treatment. The subjects were included in the SS for safety analysis.
Arm/Group | CZP 200 mg Q2W (SS) | Placebo->OL CZP (SS)
Number analyzed (Participants) | 148 | 0
µg/mL | 50.5 [48.0 to 53.0] |

5. Primary Outcome: Certolizumab Pegol Plasma Concentration at Week 2
Description: Certolizumab pegol plasma concentration was measured at Week 2, in µg/mL.
Time Frame: Week 2
Population: The SS consisted of all subjects who received at least 1 dose of study treatment. Note: No samples taken at Week 2 for the Placebo->OL CZP.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | CZP 200 mg Q2W (SS) | Placebo->OL CZP (SS)
Number analyzed (Participants) | 153 | 0
µg/mL | 36.4 [33.0 to 40.1] |

6. Primary Outcome: Certolizumab Pegol Plasma Concentration at Week 4
Description: Certolizumab pegol plasma concentration was measured at Week 4, in µg/mL.
Time Frame: Week 4
Population: The SS consisted of all subjects who received at least 1 dose of study treatment.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | CZP 200 mg Q2W (SS) | Placebo->OL CZP (SS)
Number analyzed (Participants) | 155 | 93
µg/mL | 54.6 [51.4 to 58.0] | 48.8 [42.2 to 56.4]

7. Primary Outcome: Certolizumab Pegol Plasma Concentration at Week 12
Description: Certolizumab pegol plasma concentration was measured at Week 12, in µg/mL.
Time Frame: Week 12
Population: The SS consisted of all subjects who received at least 1 dose of study treatment.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | CZP 200 mg Q2W (SS) | Placebo->OL CZP (SS)
Number analyzed (Participants) | 143 | 93
µg/mL | 29.1 [24.0 to 35.2] | 30.5 [26.4 to 35.3]

8. Primary Outcome: Certolizumab Pegol Plasma Concentration at Week 24
Description: Certolizumab pegol plasma concentration was measured at Week 24, in µg/mL.
Time Frame: Week 24
Population: The SS consisted of all subjects who received at least 1 dose of study treatment.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | CZP 200 mg Q2W (SS) | Placebo->OL CZP (SS)
Number analyzed (Participants) | 135 | 86
µg/mL | 23.5 [18.5 to 29.7] | 24.8 [20.6 to 29.9]

9. Primary Outcome: Certolizumab Pegol Plasma Concentration at Week 36
Description: Certolizumab pegol plasma concentration was measured at Week 36, in µg/mL.
Time Frame: Week 36
Population: The SS consisted of all subjects who received at least 1 dose of study treatment.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | CZP 200 mg Q2W (SS) | Placebo->OL CZP (SS)
Number analyzed (Participants) | 123 | 65
µg/mL | 24.0 [19.0 to 30.4] | 22.9 [18.3 to 28.7]

10. Primary Outcome: Certolizumab Pegol Plasma Concentration at Week 52
Description: Certolizumab pegol plasma concentration was measured at Week 52, in µg/mL.
Time Frame: Week 52
Population: The SS consisted of all subjects who received at least 1 dose of study treatment. Note: No samples taken at OL Week 52 for the Placebo->OL CZP.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | CZP 200 mg Q2W (SS) | Placebo->OL CZP (SS)
Number analyzed (Participants) | 123 | 0
µg/mL | 22.6 [17.8 to 28.6] |

11. Primary Outcome: Certolizumab Pegol Plasma Concentration at Follow-Up (FU) Visit
Description: Certolizumab pegol plasma concentration was measured at the Follow-Up Visit, in µg/mL.
  Follow-Up Visit was defined as 8 weeks after Week 52 or Withdrawal (WD) visit for subjects not participating in the Safety Follow-Up Extension (SFE) Period.
Time Frame: Follow-up Visit (up to Week 60)
Population: The SS consisted of all subjects who received at least 1 dose of study treatment. Only participants included, who had a SFU Visit at 8 weeks after Week 52/WD visit for those not participating in the SFE period.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | CZP 200 mg Q2W (SS) | Placebo->OL CZP (SS)
Number analyzed (Participants) | 17 | 10
µg/mL | 0.2 [0.1 to 0.7] | NA [NA to NA] — Values were below the level of quantification.

12. Secondary Outcome: Percentage of Subjects With Axial SpondyloArthritis International Society 40% Response Criteria (ASAS40) Response at Week 52
Description: The ASAS40 response was defined as relative improvements of at least 40% and absolute improvement of at least 2 units on a 0 to 10 Numeric Rating Scale (NRS), where 0 is "not active" and 10 is "very active" in at least 3 of the 4 domains: Patient's Global Assessment of Disease Activity (PGADA), Pain assessment (total spinal pain NRS scores), Function (Bath Ankylosing Spondylitis Functional Index (BASFI)), Inflammation (mean of Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)) questions 5 and 6 concerning morning stiffness intensity and duration) and no worsening at all in the remaining domain.
Time Frame: Week 52
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 159
percentage of subjects | 15.8 | 56.6
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); Odds ratio: CZP/Placebo and p-value were calculated using logistic regression with factors for treatment, region MRI/CRP classification; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.359, 95% CI 2-sided [4.286 to 12.636]

13. Secondary Outcome: Change From Baseline to Week 12 in the Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: The BASFI is a validated disease-specific instrument for assessing physical function. The BASFI comprises 10 items relating to the past week. The BASFI is the mean of the 10 scores such that the total score ranges from 0 (Easy) to 10 (Impossible), with lower scores indicating better physical function. The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Baseline to Week 12
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 159
scores on a scale | -0.38 (0.21) | -2.07 (0.20)
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); From an ANCOVA model including scores at Baseline, treatment group, region and MRI/CRP classification; Test type: Other; p < 0.001, ANCOVA; Difference = -1.696, 95% CI 2-sided [-2.110 to -1.282]

14. Secondary Outcome: Change From Baseline to Week 52 in the Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: as for outcome 13
Time Frame: From Baseline to Week 52
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 159
scores on a scale | -1.44 (0.30) | -3.03 (0.24)
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); From an ANCOVA model including scores at Baseline, treatment group, region and MRI/CRP classification; Test type: Other; p < 0.0001, ANCOVA; Difference = -1.585, 95% CI 2-sided [-2.132 to -1.038]

15. Secondary Outcome: Change From Baseline to Week 12 in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: The BASDAI is a validated self-reported instrument, which consists of six 10 unit horizontal Numeric Rating Scales to measure the disease activity of ankylosing spondylitis (AS) from the subject's perspective. It measures the severity of fatigue, spinal and peripheral joint pain and swelling, enthesitis, and morning stiffness (both severity and duration) over the last week. The final BASDAI scores ranges from 0 (not active) to 10 (very active), with lower scores indicating lower disease activity. The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Baseline to Week 12
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 159
scores on a scale | -0.91 (0.22) | -2.73 (0.21)
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); From an ANCOVA model including scores at Baseline, treatment group, region and MRI/CRP classification; Test type: Other; p < 0.001, ANCOVA; Difference = -1.819, 95% CI 2-sided [-2.250 to -1.388]

16. Secondary Outcome: Change From Baseline to Week 52 in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI)
Description: as for outcome 15
Time Frame: From Baseline to Week 52
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 159
scores on a scale | -2.59 (0.37) | -3.88 (0.27)
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); From an ANCOVA model including scores at Baseline, treatment group, region and MRI/CRP classification; Test type: Other; p < 0.001, ANCOVA; Difference = -1.290, 95% CI 2-sided [-1.909 to -0.672]

17. Secondary Outcome: Change From Baseline to Week 12 in Sacroiliac Spondyloarthritis Research Consortium of Canada (SI-SPARCC) Score
Description: The Spondyloarthritis Research Consortium of Canada (SPARCC) scoring method for lesions found on the Magnetic Resonance Imaging (MRI) is based on an abnormal increased signal on the Short-Tau-Inversion Recovery (STIR) sequence, representing bone marrow edema. Total Sacroiliac (SI) joint SPARCC score can range from 0 to 72 with higher scores indicating higher joint inflammation. The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Baseline to Week 12
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 159
scores on a scale | 0.200 (0.772) | -4.669 (0.770)
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); From an ANCOVA model including scores at Baseline, treatment group, region and MRI/CRP classification; Test type: Other; p < 0.001, ANCOVA; Difference = -4.8687, 95% CI 2-sided [-6.4014 to -3.3360]

18. Secondary Outcome: Number of Subjects Without Relevant Changes to Background Medication From Baseline to Week 52
Description: The number of subjects who did not have relevant changes to background medications during the study treatment period.
  A subject is without relevant changes to background medication if they do not have: the addition of a new disease-modifying antirheumatic drug (DMARD) or the change from one DMAR to another; the addition of an nonsteroidal anti-inflammatory drug (NSAID) or the change from one NSAID to another; an increased dose of chronic corticosteroids; the addition of a new chronic analgesic medication or increased dose in chronic analgesic medication; and they complete double-blind study treatment to Week 52.
Time Frame: From Baseline to Week 52
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 159
Participants | 48 | 115
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); [analysis description as in outcome 2, analysis 1]; Test type: Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.223, 95% CI 2-sided [3.800 to 10.191]

19. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) at Week 52
Description: The ASQoL score ranged from 0 to 18 with higher score indicating worse Health-Related Quality of Life (HRQoL) and 0 indicating good HRQoL. The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Baseline to Week 52
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 159
scores on a scale | -0.18 (0.04) | -0.36 (0.03)
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); From an ANCOVA model including scores at Baseline, treatment group, region and MRI/CRP classification; Test type: Other; p < 0.001, ANCOVA; Difference = -0.183, 95% CI 2-sided [-0.250 to -0.117]

20. Secondary Outcome: Change From Baseline in ASQoL at Week 1
Description: as for outcome 19
Time Frame: From Baseline to Week 1
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 150 | 147
scores on a scale | -0.03 (0.14) | -0.11 (0.21)

21. Secondary Outcome: Change From Baseline in ASQoL at Week 2
Description: as for outcome 19
Time Frame: From Baseline to Week 2
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 156
scores on a scale | -0.03 (0.15) | -0.16 (0.23)

22. Secondary Outcome: Change From Baseline in ASQoL at Week 4
Description: as for outcome 19
Time Frame: From Baseline to Week 4
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 156
scores on a scale | -0.06 (0.19) | -0.18 (0.23)

23. Secondary Outcome: Change From Baseline in ASQoL at Week 12
Description: as for outcome 19
Time Frame: From Baseline to Week 12
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 156
scores on a scale | -0.08 (0.22) | -0.28 (0.26)

24. Secondary Outcome: Change From Baseline in ASQoL at Week 24
Description: as for outcome 19
Time Frame: From Baseline to Week 24
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 156
scores on a scale | -0.09 (0.23) | -0.31 (0.27)

25. Secondary Outcome: Change From Baseline in ASQoL at Week 36
Description: as for outcome 19
Time Frame: From Baseline to Week 36
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 156
scores on a scale | -0.11 (0.23) | -0.33 (0.29)

26. Secondary Outcome: Change From Baseline in ASQoL at Week 48
Description: as for outcome 19
Time Frame: From Baseline to Week 48
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 156
scores on a scale | -0.10 (0.24) | -0.34 (0.30)

27. Secondary Outcome: Change From Baseline in Nocturnal Spinal Pain Numerical Rating Scale (NRS) at Week 52
Description: The nocturnal spinal pain experienced by subjects due to AS was measured by following question 'How much pain of your spine due to spondylitis do you have at night?'. The NRS ranged from 0 to 10, where 0 represented 'no pain' and 10 represented 'most severe pain'. The change from Baseline is calculated, a negative value indicating improvement and a positive value worsening.
Time Frame: From Baseline to Week 52
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 159
scores on a scale | -2.1 (0.5) | -4.0 (0.4)
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); From an ANCOVA model including scores at Baseline, treatment group, region and MRI/CRP classification; Test type: Other; p < 0.001, ANCOVA; Difference = -1.90, 95% CI 2-sided [-2.62 to -1.18]

28. Secondary Outcome: Number of Subjects With Anterior Uveitis (AU) or New AU Flares Through Week 52
Description: The number of subjects with AU or new AU flares during the study treatment period.
Time Frame: Throughout the study conduct (up to Week 52)
Population: The FAS consisted of all subjects in the RS who have received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (FAS) | CZP 200 mg Q2W (FAS)
Number analyzed (Participants) | 158 | 159
Participants | 8 | 4
Statistical Analysis 1: Comparison: Placebo (FAS) vs CZP 200 mg Q2W (FAS); Odds ratio: CZP/PBO and p-value were calculated using logistic regression with factors for treatment, region and MRI/CRP classification; Test type: Other; p = 0.247, Regression, Logistic; Odds Ratio (OR) = 0.484, 95% CI 2-sided [0.142 to 1.653]

29. Secondary Outcome: Percentage of Subjects With Treatment-Emergent Adverse Events (TEAEs) During the Study
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From Baseline up to the End of Safety Follow-up Extension Period (up to Week 156)
Population: The SS consisted of all subjects who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of subjects
Groups:
- CZP->OL CZP (SS): Subset of subjects from the CZP 200 mg Q2W group, who discontinued the CZP double-blind treatment and entered the CZP open-label treatment. The subjects were included in the SS for safety analysis.
- SFE OL CZP 200 mg Q2W (SS): Subjects who completed Double-Blind Period received CZP 200 mg at Week 52, 54 and 56 to maintain the blinding and who completed the Week 52 Visit on placebo treatment received loading doses of CZP 400 mg at these visits. Subjects who completed the Week 52 Visit on CZP treatment received 1 injection of CZP 200 mg and 1 injection of placebo at these visits to continue their previous CZP treatment regimen and subjects who discontinued from Double-Blind Period and entered OL CZP treatment continued their OL CZP treatment regimen during SFE Period. The subjects were included in the SS for safety analysis. Subjects received CZP 200 mg Q2W for up to 2 years during the SFE Period. An additional signed informed consent for the SFE was a pre-requisite For the additional milestone one (Received OL CZP; Completed Week 52 without starting SFE) reported in Double-Blind Period (Week 0 -52).
Arm/Group | Placebo (SS) | CZP 200 mg Q2W (SS) | Placebo->OL CZP (SS) | CZP->OL CZP (SS) | SFE OL CZP 200 mg Q2W (SS)
Number analyzed (Participants) | 158 | 159 | 96 | 20 | 243
percentage of subjects | 63.9 | 75.5 | 59.4 | 65.0 | 61.3

30. Secondary Outcome: Percentage of Subjects With Serious Adverse Events (SAEs) During the Study
Description: A serious adverse event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Is an infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above.
Time Frame: From Baseline up to the End of Safety Follow-up Extension Period (up to Week 156)
Population: The SS consisted of all subjects who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo (SS) | CZP 200 mg Q2W (SS) | Placebo->OL CZP (SS) | CZP->OL CZP (SS) | SFE OL CZP 200 mg Q2W (SS)
Number analyzed (Participants) | 158 | 159 | 96 | 20 | 243
percentage of subjects | 2.5 | 5.0 | 3.1 | 5.0 | 6.2

31. Secondary Outcome: Percentage of Subjects With Adverse Events Leading to Withdrawal From Investigational Medicinal Product (IMP) During the Study
Description: as for outcome 29
Time Frame: From Baseline up to the End of Safety Follow-up Extension Period (up to Week 156)
Population: The SS consisted of all subjects who received at least 1 dose of study treatment.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo (SS) | CZP 200 mg Q2W (SS) | Placebo->OL CZP (SS) | CZP->OL CZP (SS) | SFE OL CZP 200 mg Q2W (SS)
Number analyzed (Participants) | 158 | 159 | 96 | 20 | 243
percentage of subjects | 1.9 | 1.9 | 3.1 | 0 | 2.5

ADVERSE EVENTS:
Time Frame: From Baseline up to the End of Safety Follow-up Extension Period (up to Week 156)
Description: Adverse events were recorded for all subjects, including those who discontinued the blinded treatment and entered the open-label treatment with CZP (OL). Based on this the following groups were generated: Placebo, Placebo-> OL CZP, CZP, CZP->OL CZP and OL CZP during SFE Period for all subjects entering the SFE Period.
Arm/Group | Placebo (SS) | CZP 200 mg Q2W (SS) | Placebo->OL CZP (SS) | CZP->OL CZP (SS) | SFE OL CZP 200 mg Q2W (SS)
All-Cause Mortality (participants affected / at risk) | 0/158 | 0/159 | 0/96 | 0/20 | 0/243
Serious Adverse Events (participants affected / at risk) | 4/158 | 8/159 | 3/96 | 1/20 | 15/243
Other Adverse Events (participants affected / at risk) | 59/158 | 75/159 | 27/96 | 7/20 | 69/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) (N=158) | CZP 200 mg Q2W (SS) (N=159) | Placebo->OL CZP (SS) (N=96) | CZP->OL CZP (SS) (N=20) | SFE OL CZP 200 mg Q2W (SS) (N=243)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuroborreliosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervix neoplasms (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrosalpinx (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian enlargement (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (SS) (N=158) | CZP 200 mg Q2W (SS) (N=159) | Placebo->OL CZP (SS) (N=96) | CZP->OL CZP (SS) (N=20) | SFE OL CZP 200 mg Q2W (SS) (N=243)
Diarrhoea (Gastrointestinal disorders) | 10 (10) | 8 (11) | 1 (1) | 0 (0) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 16 (23) | 30 (38) | 10 (14) | 4 (5) | 21 (31)
Nasopharyngitis (Infections and infestations) | 13 (17) | 21 (24) | 10 (13) | 0 (0) | 26 (33)
Bronchitis (Infections and infestations) | 5 (5) | 8 (9) | 5 (5) | 0 (0) | 10 (11)
Blood creatine phosphokinase increased (Investigations) | 4 (4) | 8 (9) | 1 (1) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 9 (12) | 2 (2) | 2 (2) | 6 (6)
Axial spondyloarthritis (Musculoskeletal and connective tissue disorders) | 12 (13) | 11 (13) | 0 (0) | 0 (0) | 5 (5)
Headache (Nervous system disorders) | 7 (9) | 11 (15) | 0 (0) | 3 (3) | 9 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 6 (6) | 2 (2) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT02552212/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT02552212/SAP_002.pdf